CLINICAL TRIAL: NCT01493245
Title: A Phase 3 Study of JNS020QD in Patients With Chronic Pain
Brief Title: A Study of JNS020QD in Patients With Chronic Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR018745; JNS020QD-JPN-N04 (Other: Janssen Pharmaceutical K.K., Japan)
Record Dates: First submitted 2011-12-08; First posted 2011-12-15 (Estimated); Last update posted 2014-03-24 (Estimated); Status verified 2014-03

CONDITIONS: Chronic Pain
Keywords: Chronic Pain; JNS020QD; Fentanyl; Opioid analgesics
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- JNS020QD (Experimental)
  Interventions: Drug: JNS020QD

INTERVENTIONS:
Drug: JNS020QD — During weeks 1-3, initial doses of 0.84 mg, 1.7 mg, 3.4 mg, or 5 mg can be increased until individual optimal dose (up to maximum 20.1 mg) is determined. The optimal dose will be administered during the maintenance period (1 week), followed by a long-term treatment (48 weeks) period, where the dose will be adjusted (escalated or reduced) in consideration of the efficacy of the study, and the condition of adverse events. The patches are applied on the skin and exchanged daily (every 24 hours) for consecutive 52 weeks.

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of JNS020QD in patients with moderate to severe chronic pain who switched from opioid analgesics, as well as the safety and efficacy of long-term treatment (52 weeks) after switching to JNS020QD.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the efficacy and safety of JNS020QD in patients with moderate to severe chronic pain who are switching from opioid analgesics. It will also evaluate the safety and efficacy of long-term treatment (52 weeks) after switching to JNS020QD. The study will enroll patients with moderate to severe chronic pain which is adequately controlled with a regular treatment with an opioid analgesic agent other than the study drug because these patients are considered appropriate to investigate the conversion ratio in switching from JNS020QD to other opioid analgesics, and to evaluate the efficacy and safety of the study drug. This is an open-label (all people know the identity of the intervention), uncontrolled (the study does not involve a control treatment), multicenter study. This study consists of Screening period (1 to 2 weeks), Period I (3-week titration period+ 1-week maintenance period), Period II (48 weeks long-term treatment period), tapering period (if required, 0 to 6 weeks), and follow-up period (1 week). JNS020QD is a transdermal system in which fentanyl base is incorporated directly into a single layer of pressure-sensitive high polymerized adhesive, and is changed once a day (every 24 hours). JNS020QD is available in 5 formulations containing fentanyl 0.84 mg, 1.7 mg, 3.4 mg, 5 mg, or 6.7 mg per system.. The study drug patch will be applied to the breast, abdomen, upper arm, femoral region, etc. exchanged daily and for consecutive 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Chronic pain that requires opioid analgesics and that has persisted for 12 weeks or longer before giving the consent
* Patients who received any of the following opioid analgesics at a stable dose for the treatment of chronic pain for 7 days or longer before giving the consent (excluding rescue dose): oral codeine phosphate; oral morphine hydrochloride; fentanyl transdermal; combination tablet of tramadol hydrochloride and acetaminophen; buprenorphine transdermal patch
* Patients who received 2 or less rescue doses per day during the 7 days before giving consent
* Patients whose mean pain intensity throughout the day of giving the consent is 45 mm or less on the visual analogue scale (VAS)
* Male and female patients surgically sterile, abstinent, or practicing an effective method of birth control. Female patients have a negative pregnancy test result at screening. Male patients cannot donate sperm during the study and for 3 months after receiving the last dose of study drug

Exclusion Criteria:

* Other painful conditions which may interfere with the efficacy evaluation (eg bone fracture, rheumatoid arthritis)
* Major surgery within 30 days before screening, or not fully recovered from surgery, or planned surgery during the time of the study
* Pain that is considered mainly psychogenic
* Uncontrolled/clinically significant arrhythmia
* Hepatic function disorder such as fulminant hepatitis and hepatic cirrhosis, or renal impairment such as nephritic syndrome, acute or chronic renal failure
* Any other condition that, in the opinion of the investigator, would compromise the best interest of the patient or that could prevent, limit, or confound the protocol-specified assessments

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2011-10; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who maintained the adequate analgesia | At Week 4
  Criteria for maintenance of adequate analgesia is defined as: 1) The daily dose of the study drug is constant during the 7 days in the maintenance period before completion of the maintenance period; 2) Change in Visual Analogue Scale (VAS) mean values from baseline to endpoint is ≤+15 mm; 3) Frequency of daily rescue doses during the 7 days in the maintenance period is ≤ 2 doses, and the change in the mean frequency of daily rescue dose from the baseline to endpoint is ≤+1.0 dose.

SECONDARY OUTCOMES:
Proportion of patients who achieve dose-adjustment | Days 19-21
  Criteria for achievement of dose-adjustment is defined as: 1) The daily dose of the study drug is constant during the 3 days before completion of the titration period; 2) Change in Visual Analogue Scale (VAS) mean values from baseline to endpoint is ≤+15 mm; 3) Frequency of daily rescue doses during the 3 days in the titration period is ≤2 doses; 4) daily doses of the study drug during the titration period does not exceed the maximum doses stipulated by the investigators.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K., Japan Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (18):
- Japan (18):
  - Asahikawa
  - Chiba
  - Isesaki
  - Izumo
  - Kawasaki
  - Kobe
  - Matsumoto
  - Nishinomiya
  - Ohtsu
  - Okayama
  - Osaka
  - Saga
  - Sagamihara
  - Sapporo
  - Sendai
  - Toyama
  - Yamagata
  - Yamaguchi

REFERENCES:
- See also: A Phase 3 Study of JNS020QD in Patients with Chronic Pain — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=3333&filename=CR018745_CSR.pdf